CLINICAL TRIAL: NCT03288636
Title: A Phase I Study to Assess the Pharmacokinetics and Safety of Single Dose of Ravidasvir and Danoprevir/r and Repeated Doses of Ravidasvir in Combination With Danoprevir/r in Healthy Volunteers.
Brief Title: Pharmacokinetics and Safety of ASC16 Tablets in Healthy Volunteers in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC-ASC16-I-CTP-02
Record Dates: First submitted 2017-08-09; First posted 2017-09-20 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-10

CONDITIONS: HCV
MeSH Terms: interventions — danoprevir; Ritonavir; ravidasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): PKGroup:
  Ravidasvir + Danoprevir/ Ritonavir
  Interventions: Drug: Danoprevir; Drug: Ritonavir; Drug: Ravidasvir
- Placebo (Placebo Comparator): Placebo Group:
  Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danoprevir — Danoprevir tablet administered orally 100mg QD on day 7 and 13, 100mg BID on day 14-22, 100mg QD on day 23
  Arms: Experimental
Drug: Ritonavir — Ritonavir tablet administered orally 100mg QD on day 7 and 13, 100mg BID on day 14-22, 100mg QD on day 23
  Arms: Experimental
Drug: Ravidasvir — Ravidasvir tablet administered orally 200mg QD on day 1, 13 - 23
  Other Names: ASC16(RDV)
  Arms: Experimental
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the Pharmacokinetics and Safety of single dose of Ravidasvir and Danoprevir/r and repeated doses of Ravidasvir in combination with Danoprevir/r in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years old;
* Male body weight not less than 50kg; Female body weight not less than 45kg; BMI in the range of 19~28kg/m2
* Healthy men or women based on history, physical examination, laboratory examination and ECG.
* Female subjects should be surgically sterilized (bilateral tubal ligation, bilateral ovariectomy or hysterectomy); or are willing to use at least one of the following contraceptive methods within 30 days of the first administration of the study drug until the last administration: I Male partner vas deferens ligation; II. Non-hormonal contraceptive methods: intrauterine contraceptives, condoms, contraceptive sponges, septa, vaginal ring containing sizing gel or cream.
* Male subjects should be surgically sterilized; or are willing to use at least one of the following contraceptive methods within 30 days from the first administration of the study to the last administration: I. Female partners abstinence during the study period (including no donation): II. Compounds use hormonal contraceptives (oral, vaginal, parenteral or transdermal); III. Subjects and / or their female partners use non-hormonal contraceptive methods: condoms, contraceptive sponges, membranes, intrauterine devices, Fine gel or cream of the vaginal ring.
* If female, the pregnancy test result should be negative during the screening period.
* Voluntary to sign the informed consent.

Exclusion Criteria:

* History or presence of cardiovascular disease, respiratory disease, endocrine and metabolic system disease, urinary system, digestive system, hematological system diseases, nervous system or Psychiatric diseases, and acute or chronic infectious disease and malignant tumor.
* A history of drug or food allergy.
* Positive test in any of the HBsAg、HCV Ab、HIV Ab and Syphilis Ab.
* Any of the AST、ALT、ALP、TBIL and DBIL exceed the upper limits of normal, or other laboratory test results exceeding the normal range and judged by the investigator to be clinically significant.
* History of gastrointestinal surgery, trunk vagotomy, intestinal excision or any other surgeries that could disturb gastrointestinal motility and PH absorption.
* Female who were during pregnancy, breastfeeding, period and unwilling to take reliable birth control method.
* Female partners were fertile and unwilling to take reliable contraceptive measures.
* Others as specified in the detailed protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 40 days
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Zhejiang province, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu G, Zhou H, Wu J, Lv D, Wu L, Zhai Y, Lin M, Wu JJ, Shentu J. Pharmacokinetics, Safety, and Tolerability of Ravidasvir, with and without Danoprevir/Ritonavir, in Healthy Subjects. Antimicrob Agents Chemother. 2021 Sep 17;65(10):e0060021. doi: 10.1128/AAC.00600-21. Epub 2021 Jul 12. PMID 34252301